CLINICAL TRIAL: NCT05408156
Title: Effects of Customized Insoles for Individuals With Symptomatic Hallux Valgus: Protocol for a Sham-controlled Randomized Trial
Brief Title: Effects of Customized Insoles for Individuals With Symptomatic Hallux Valgus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Marcelo Cardoso de Souza, PT, PhD., Adjunct Professor, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UFRNHáluxValgus
Record Dates: First submitted 2022-05-26; First posted 2022-06-07 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Hallux Valgus; Foot Diseases; Foot Deformities
Keywords: hallux valgus; insoles; pain
MeSH Terms: conditions — Hallux Valgus; Foot Diseases; Foot Deformities; Pain | interventions — Foot Orthoses

STUDY DESIGN:
Intervention Model Description: Customized insoles group and Sham Insoles Group
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All assessments will be performed by researcher A, who will not be involved with the interventions and will remain blind to the identification of groups. The results of the evaluations will be delivered to researcher C, a researcher with experience in making the insoles, so that they can be made. GPC participants will receive the insoles according to the assessment measurements, five days after the assessment start date.
  Each participant will remain identified by numbers and not names. Participants will be informed about the purpose of the study to compare the two interventions using customized insoles. In order not to compromise the blinding of the study, all participants will be submitted to the same evaluation before the production and delivery of the insoles. When the insoles are ready, participants will be scheduled for removal at different times, avoiding possible meetings or exchange of information.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Customized insoles group (Experimental): The participant allocated in the CIG will receive a semi-flexible non-moulded insole with a 2.5mm coverage with Shore A 28, a 5mm retrocapital bar with a Shore A 22 and a 2mm infracapital bar of the first metatarsal with a Shore A 35, produced in acetate. -ethylene vinyl (EVA) and manufactured by researcher C. The insole will be used on both feet to maintain symmetry between the limbs and generate greater comfort, since this will not be a corrective intervention.
  Interventions: Other: Insoles
- Sham Insoles Group (Sham Comparator): The SIG will receive the same unmolded insole with a semi-flexible base and 2.5mm coverage with Shore A 28, but without the bars used in the intervention group.
  Interventions: Other: Insoles

INTERVENTIONS:
Other: Insoles — semi-flexible non-moulded insole with a 2.5mm coverage with Shore A 28, a 5mm retrocapital bar with a Shore A 22 and a 2mm infracapital bar of the first metatarsal with a Shore A 35, produced in acetate ethylene vinyl (EVA)

SUMMARY:
Hallux valgus is one of the most common forefoot deformities. Its prevalence increases with age, representing approximately 23% in adulthood, being more common in females. Some studies indicate that the use of the insole associated with the finger separator promotes pain relief and that this may be related to better alignment of the hallux. However, there is still no consensus about the ideal insole or how long it should be used to relieve pain or improve function in patients with hallux valgus. Therefore, the objective of this study will be to evaluate the effect of the customized insole on pain and function of individuals with symptomatic hallux valgus.

DETAILED DESCRIPTION:
This is a protocol for a randomized, controlled, blinded clinical trial. Eighty participants with hallux valgus pain will be evaluated and randomized into two intervention groups (40 per group): customized insole group or sham insole group. Assessments will be performed at baseline (T0), after six weeks (T6) and twelve weeks (T12) of insoles use, in addition to the follow-up that will be performed four weeks after the end of the intervention (T16). The primary outcome will be pain, assessed by the Numerical Pain Scale and the secondary outcome will be foot functionality, assessed by the Foot Function Index questionnaire. Statistical analysis: For normal data, analysis of variance with a mixed design will be considered, and for non-normal data, the Friedman test will be used, in addition to the interaction of time per group and intergroup and intragroup differences. The Bonferroni test will be performed in post hoc analyses. Intent-to-treat analysis will be used. A significance level of 5% and CI 95% will be adopted for all statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both sexes aged over 18 years;
* Presence of mild to moderate hallux valgus, according to the Manchester scale;
* Presenting no hallux with intensity greater than or equal to 3 points up to 8 points, according to the Numerical Pain Scale (END);
* Be available to actively use the insole for at least 4 hours/day;
* Commitment to wear closed shoes, for example (sneakers, shoes used by the patient, due to: wide toe cap and heel height of 2 to 3 cm) during the study.

Exclusion Criteria:

* Being in physical therapy treatment for hallux valgus concomitantly with the research;
* Previous hallux valgus surgeries performed in the last 5 years;
* Presence of foot wounds and wounds, dislocations or metatarsophalangeal fractures in the foot with HV, in the last 5 years
* Presence of diseases such as rheumatoid arthritis, decompensated diabetes, gout, neurodegenerative diseases;
* Cognitive and mental disorder being unable to respond; those related to the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Numerical Pain Scale (END) | baseline, 6 weeks, 12 weeks, 16 weeks
  Pain intensity will be assessed using the Numerical Pain Scale (END), in which individuals will classify their pain on a numerical scale from 0 to 10 points. This scale will be positioned in front of the participant and will vary from zero to ten points, with zero being the complete absence of pain and ten being the worst pain imaginable by the individual. The quantification of pain intensity will be evaluated at the first steps in the morning and throughout the day.

SECONDARY OUTCOMES:
Change in Foot Function Index (FFI) | baseline, 6 weeks, 12 weeks, 16 weeks
  Foot functionality will be measured by the Foot Function Index (FFI) questionnaire, which is capable of measuring the impact of foot pathologies related to pain, disability and activity restriction on the function. It consists of 23 items grouped into three subscales, five items related to disability, nine items related to pain and nine items about activity limitation32. The final result will be the average of all domains (the values are added and divided by three). Results can range from 0 to 100% and are directly proportional to the functional impairment of the foot.
Change in Treatment expectation | baseline
  Treatment expectations will be assessed using a 5-point Likert scale. The following will be asked to participants at T0: "Do you think that by using customized insoles, you will: 1- get much worse, 2 - get worse, 3 - no changes, 4 - improve, or 5 - greatly improve?"
Change in Self-assessment of treatment | 16 weeks
  A 5-point Likert scale will be used to assess satisfaction with the intervention. Participants will be asked the following question: "How are you feeling after using the insoles?: 1- much worse, 2 - worse, 3 - no changes, 4 - better, or 5 - much better."
  A 5-point Likert scale will be used to assess satisfaction with the intervention. Participants will be asked the following question: "How are you feeling after using the insoles?: 1- much worse, 2 - worse, 3 - no changes, 4 - better, or 5 - much better."
Change in Blinding test | 16 weeks
  Participants will be asked which group they believed they were allocated: CIG or SIG. This strategy has been recommended at the end of clinical trials to test whether the blinding strategy adopted was effective Blinding test
Change in Hours of insole use | 16 weeks
  Participants of both groups will receive an insole control diary to register the number of hours per day spent with the insole. Participants should keep the diary for 12 weeks and return it to researchers at T12. Monitoring and motivation will be performed via telephone or WhatsApp messages to prevent participants from forgetting to use the insole

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo C de Souza, PT, PhD, Principal Investigator — Universidade Federal do Rio Grande do Norte
Locations (1):
- Marcelo Cardoso de Souza, Natal, Rio Grande do Norte, Brazil

IPD SHARING:
Plan to Share IPD: No
Participant data (IPD) will not be available to other investigators

REFERENCES:
- [Result] Costa ARA, de Almeida Silva HJ, Mendes AAMT, Scattone Silva R, de Almeida Lins CA, de Souza MC. Effects of insoles adapted in flip-flop sandals in people with plantar fasciopathy: a randomized, double-blind clinical, controlled study. Clin Rehabil. 2020 Mar;34(3):334-344. doi: 10.1177/0269215519893104. Epub 2019 Dec 6. PMID 31808352
- [Derived] Cavalcanti RR, Mendes AAMT, Barbosa GM, de Souza MC. Effects of custom insoles for symptomatic hallux valgus: protocol for a sham-controlled randomised trial. BMJ Open. 2023 Jul 3;13(7):e069872. doi: 10.1136/bmjopen-2022-069872. PMID 37400239